CLINICAL TRIAL: NCT04701528
Title: An Open-Label Study Evaluating Anti-Viral Effects of Voclosporin in SARS-CoV-2 Positive Kidney Transplant Recipients - the VOCOVID Study
Brief Title: Anti-Viral Effects of Voclosporin in COVID-19 Positive Kidney Transplant Recipients
Acronym: VOCOVID
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Leiden University Medical Center (Other)
Collaborators: Aurinia Pharmaceuticals Inc. (Industry)
Responsible Party: Principal Investigator, Y.K.Onno Teng, Dr. Y.K.O. Teng, MD, PhD, Leiden University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL73762.058.20
Record Dates: First submitted 2020-10-27; First posted 2021-01-08 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: Covid19; Kidney Transplant Infection
MeSH Terms: conditions — COVID-19 | interventions — voclosporin; Specimen Handling; N-acetyltalosaminuronic acid; Tacrolimus

STUDY DESIGN:
Intervention Model Description: single-center, proof-of-concept
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Voclosporin (VCS) (Experimental): Prior to or at study entry, subjects are reduced in their standard immunosuppressive therapy to dual therapy with prednisone and tacrolimus according to current local guidelines.
  In the experimental arm tacrolimus is switched to voclosporin 6 capsules (of 7.9 mg each) BID for a treatment period of minimal 56 days with a possible extension up to 1 year.
  Safety drug monitoring will take place during the study to ensure that VCS trough levels are maintained between 30-60 ng/mL. If trough levels are not within these levels, dose adjustments will take place.
  Interventions: Drug: Voclosporin
- Tacrolimus (TAC) (Active Comparator): Prior to or at study entry, subjects are reduced in their standard immunosuppressive therapy to dual therapy with prednisone and tacrolimus according to current local guidelines.
  In the Active comparator arm tacrolimus dosage is maintained.
  Safety drug monitoring will take place during the study to ensure that TAC trough levels are maintained between 3-7 ng/ml. If trough levels are not within these levels, dose adjustments will take place.
  Interventions: Drug: Tacrolimus

INTERVENTIONS:
Drug: Voclosporin — Temporarily switching of tacrolimus maintenance immunosuppression to voclosporin maintenance immunosuppression with possible additional anti-viral activity
  Other Names: Specimen collection for Nuclear acid testing (NAT) on SARS-CoV-2
  Arms: Voclosporin (VCS)
Drug: Tacrolimus — Comparator
  Other Names: Specimen collection for Nuclear acid testing (NAT) on SARS-CoV-2
  Arms: Tacrolimus (TAC)

SUMMARY:
An open-label, 56 day, single-center, exploratory, proof-of-concept study of the anti-viral effect of voclosporin (VCS) with an extended safety follow-up, up to 1 year. Study population are adult KTRs with positive SARS-CoV-2 infection with mild to moderate symptoms. At study entry, subjects are on standard therapy of dual immunosuppressive treatment of prednisone and tacrolimus (TAC), following randomization, 10 out of 20 subjects will remain on this therapy for the duration of the study, while the other 10 subjects will switch to VCS.

DETAILED DESCRIPTION:
Calcineurin inhibitors (CNIs) are general immunosuppressive agents commonly used in the setting of transplantation to prevent solid organ rejection. CNIs form the cornerstone of immunosuppressive treatment in kidney transplant recipients (KTRs) including the 1st generation CNI Cyclosporin-A (CsA) and the most commonly employed 2nd generation CNI tacrolimus (TAC). It is of interest that CNIs, especially CsA, also exert anti-viral effects in addition to immunosuppressive effects. Common side effects of CNIs are hypertension, new-onset diabetes, renal insufficiency and neurotoxicity. Therefore, in the recent decennium, efforts have been directed at developing a novel CNI, voclosporin (VCS), that has improved pharmacodynamic (PD) and pharmacokinetic (PK) attributes with respect to calcineurin inhibition as well as an improved safety profile to common side effects. VCS has been extensively studied in KTRs demonstrating equivalent efficacy to TAC with respect to prevention of rejection while showing a reduction in CNI-related toxicity. Most recently, VCS as a component of multitargeted therapy demonstrated superior efficacy compared to standard of care in lupus nephritis (LN) patients.

In 2011, a pivotal study from Leiden University Medical Center (LUMC) demonstrated in vitro anti-viral effect of CsA on Severe Acute Respiratory Syndrome Coronavirus-1 (SARS-CoV-1). Subsequently, VCS has been shown to have a more potent anti-viral effect on norovirus compared to CsA. The anti-viral effects of CNIs have a different mechanism of inhibition in each virus but mainly through inhibiting cyclophilins, an essential protein for viral replication. The SARS-CoV-1 interacts with human cyclophilins, however the role of these proteins in infection remains elusive. Different reports stablished interactions between nsp1 or nucleocapsid proteins with Cyps and hypothesize its influence in viral replication and viral entry. Unlike VCS and CsA, TAC binds to FK binding proteins rather than cyclophilin A (CypA). Given the current COVID-19 pandemic, the LUMC has very recently demonstrated anti-viral effects of CNIs on SARS-CoV-2 infected cells in vitro: a 2-log reduction of SARS-CoV-2 viral titers in Calu-3 2B4 bronchial cell cultures was observed when incubated with ~3 μM VCS compared to 25μM CsA and 25μM TAC. In each experiment Remdesivir was taken as positive control as it inhibits viral replication by >4log at 10 μM concentration. As such, VCS becomes an attractive and potentially feasible CNI to use or switch to in COVID-19 infected KTRs who are already using CNIs as part of their chronic immunosuppressive therapy.

Because subjects will be randomized to either VCS or TAC as immunosuppressive agent during COVID-19 infection, the burden of the study is two-fold: first, subjects will need to switch to a novel CNI which intrinsically will harbour an uncertainty. However, from a clinical point-of-view VCS is proven equivalent to TAC with respect to organ rejection and safety monitoring of adequate drug levels is incorporated in the study. Secondly, subjects will need to agree to self-assessments including monitoring of vital signs and collection of saliva samples and a throat swab in the first 56 days. We believe that it is actually in the interest of subjects to undergo this intensive monitoring because current standard practice is for KTRs with mild symptoms to not be hospitalized and stay at home until recovery without further monitoring. In addition, blood sampling (10 x 38.5 mL), urine sampling and additional hospital visits will take place which are outside of normal clinical practice.

The potential advantage of the study to KTRs is that VCS may lead to a quicker reduction of SARS-CoV-2 viral load and quicker relief of symptoms. Altogether, we believe the burden of the study is minimal and outweighed by the potential benefit of the treatment on COVID-19 infection.

ELIGIBILITY:
Inclusion Criteria:

1. Provide written informed consent.
2. Male or female subjects with a minimum age of 18 years at Visit 1.
3. Subjects with a stable kidney transplant taking TAC and a confirmed diagnosis of SARS-CoV-2 by nuclear acid testing, with mild-to-moderate symptoms.
4. Patients with mild-to-moderate disease symptoms in which mild disease is defined by non-hospitalized patients without oxygen need and moderate disease symptoms are defined by hospitalization to a nursing ward with the need of oxygen therapy.
5. Women of childbearing potential must have a negative pregnancy test at baseline. Two effective forms of contraception must be used simultaneously unless abstinence is the chosen method. Subjects must use effective contraception during the study.

Exclusion Criteria:

1. Subjects unable or unwilling to give written informed consent and/or to comply with study procedures.
2. Any known hypersensitivity or contraindication to CNIs, especially CsA, or components of any cyclosporine drug product.
3. Current or medical history of:

   * Congenital immunodeficiency.
   * Severe, known, active viral infections, excluding SARS-CoV-2, within 3 months of baseline (e.g., cytomegalovirus, hepatitis B virus, hepatitis C virus or HIV) that are deemed to interfere with study assessments or outcome according to Investigator's judgement.
4. Severe symptoms resulting from SARS-CoV-2 infection defined by requiring admittance to a medium or high care unit with the need for positive pressure ventilation at baseline.
5. Other major physical or psychiatric illness or major traumatic injury or any other medical condition associated with increased risk to the subject or that may affect study conduct or interfere with study assessments or outcome according to Investigator's judgement.
6. Subjects who are pregnant, breast feeding or, if of childbearing potential, not using adequate contraceptive precautions.
7. Participation in another interventional clinical study within 4 weeks prior to baseline and/or receipt of investigational drugs within 4 weeks or 5 half-lives of the drug (whichever is longer) prior to baseline.
8. Subjects less than 3 months post-transplant.
9. Subjects with documented organ rejection within the past 3 months.
10. Subjects with a documented estimated glomerular filtration rate (eGFR) <15 ml/min within the previous 3 months prior to screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-11-15 (Actual); Primary Completion 2022-03-25 (Actual); Study Completion 2022-10-25 (Actual)

PRIMARY OUTCOMES:
Time to viral clearance of SARS-CoV-2 | Day 56
  measured by first negative reverse transcription quantitative polymerase chain reaction (RT-qPCR) with a CT value of >37 over 56 days

SECONDARY OUTCOMES:
Time to 2 consecutive negative RT-qPCR tests with CT-value >37 | Day 56
  negative test is defined as a CT-value above 37
Time to reduction in viral load | Day 56
  below 3 log copies
Time to 2 consecutive negative RT-qPCR tests with CT-value >24 | Day 56
  negative test is defined as a CT-value above 24
Time to clinical recovery | Day 56
  defined as free of symptoms for five days or more
Time to clinical symptom relief | Day 56
  defined as free of symptoms for one day or more
Time to hospital discharge | Day 56
  for hospitalized subjects
Occurrence of treatment failures | Day 56
  Worsening of COVID infection requiring hospitalization for non-hospitalized subjects OR Worsening of COVID infection for hospitalized subjects requiring admittance to the ICU or death

CONTACTS AND LOCATIONS:
Overall Officials: Y.K.O. Teng, MD, PhD, Principal Investigator — Leiden University Medical Center
Locations (1):
- Leiden University Medical Center, Leiden, Netherlands

IPD SHARING:
Plan to Share IPD: No